CLINICAL TRIAL: NCT03282019
Title: Efficacy and Safety of Long-term High-flow Nasal Cannula Oxygen Therapy in Stable COPD Patients with Home Oxygen Therapy (HOT): a Multicenter, Prospective, Randomized Controlled Study
Brief Title: Study of Long-term HFNC for COPD Patients with HOT
Acronym: FLOCOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Kobe City Medical Center General Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRIRES1668; UMIN000028581 (Registry Identifier: UMIN-CTR)
Record Dates: First submitted 2017-09-07; First posted 2017-09-13 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2021-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: myAIRVO2; high-flow nasal cannula therapy; home oxygen therapy; HOT; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A(myAIRVO2® + HOT) (Experimental): Subjects receive following protocol treatment; Home oxygen therapy (HOT) plus nocturnal high-flow nasal cannula therapy with the myAIRVO2 within 52weeks.
  Interventions: Device: High-flow nasal cannula therapy; Device: Home oxygen therapy (HOT)
- Arm B(HOT) (Active Comparator): Subjects receive following protocol treatment; Home oxygen therapy (HOT) only within 52weeks.
  Interventions: Device: Home oxygen therapy (HOT)

INTERVENTIONS:
Device: High-flow nasal cannula therapy — Subjects will receive nocturnal high-flow nasal cannula therapy with the myAIRVO2®, in addition to their current Home oxygen therapy (HOT). The myAIRVO2® is used for at least 4 hours per day with flow rates in the range 30-40 L/min. The investigator can adjust the nocturnal oxygen flow rates to keep SpO2 88-92% stably. If the subjects report discomfort, the investigator can adjust the flow rates in the range at least 20 L/min.
  Other Names: myAIRVO2®
  Arms: Arm A(myAIRVO2® + HOT)
Device: Home oxygen therapy (HOT) — All subjects will continue their current Home oxygen therapy (HOT) which kept original usage conditions at the time of enrollment throughout the entire duration of the study regardless of treatment arm assignment.

SUMMARY:
This is a prospective, randomized parallel study for evaluation of the efficacy and safety of long-term nocturnal high-flow nasal cannula therapy (HFNC: with the myAIRVO2 as HFNC in this study) in stable COPD patients with the global initiative for chronic obstructive lung disease (GOLD) stage 2-4, PaCO2 >= 45 Torr and hypercapnia who require home oxygen therapy (HOT) using COPD exacerbation (Moderate or Severe).

DETAILED DESCRIPTION:
An abroad study of the stable COPD patients was reported that HFNC usage decreased the frequency of COPD exacerbation.

In addition, the result of the pilot study (NCT02545855) of the stable COPD patient in Japan is indicated that HOT with HFNC improved their QOL and PaCO2 by comparing to HOT only.

Therefore, this study is planned to indicate the efficacy of HFNC which can increase the ventilation efficiency and have the function of heated humidification, by comparing HOT with HFNC to HOT only.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are diagnosed with the global initiative on obstructive lung disease (GOLD) stage 2-4 COPD.
2. Patients who have received nocturnal HOT 16 hours or more per day for 1 month or more at the time of the informed consent.
3. Patients with PaCO2 >= 45 Torr and pH >= 7.35 at screening.
4. Patients with COPD exacerbation (Moderate or Severe; judged by the investigators) within the past 1 year prior to the informed consent.
5. Patients who are more than 40 years old at the time of the informed consent.
6. Patients who agree to participate in the study with the written informed consent.

Exclusion Criteria:

1. Patients with severe kidney, liver or cardiovascular disease.
2. Patients with active malignant tumor.
3. Patients with acute disease.
4. Patients who are diagnosed with asthma. (Excluding COPD patients with history of asthma).
5. Patients who have any history of obstructive sleep apnea syndrome (OSAS) or are highly-suspected cases in the clinical. (Excluding patients who are denied the diagnosis of OSAS by the result of overnight polysomnography.)
6. Patients with diseases that affecting the efficacy endpoints (for example: active pulmonary infection, clinically significant pulmonary fibrosis and bronchiectasis, α-1-antitrypsin deficiency etc.,) and are regarded as inadequate for the study by the investigators.
7. Patients who have experienced a COPD exacerbation (any Severity: judged by the investigators) within the past 4 weeks prior to the informed consent.
8. Patients who are receiving nocturnal noninvasive positive pressure ventilation (NPPV), or who had been received it within 4 weeks prior to the informed consent.
9. Patients who have used HFNC at home within the past 1 year prior to the informed consent, or are using any HFNC. (Excluding patients who used HFNC during hospitalization due to acute respiratory failure within 1 year prior to the informed consent.)
10. Patients with history of tracheotomy, severe pharyngeal surgery or severe nasal cavity surgery within the past 6 months prior to the informed consent.
11. Patients who are pregnant.
12. Patients with cognitive impairment or mental disorder who are regarded as inadequate to evaluate for the study by the investigators.
13. Patients who are regarded as being unable to operate the myAIRVO2 adequately at home by the investigators.
14. Patients who have participated in the other study at the time of the informed consent, or will participate in the other study.
15. Any other cases who are regarded as inadequate for the study enrollment by the investigators.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Frequency (the number of occurrences per year) of COPD exacerbation (Moderate or Severe) | 52weeks
  COPD exacerbation will be assessed by the disease diary which is kept by each patient within the term of intervention.

SECONDARY OUTCOMES:
Term from enrollment to the date of first COPD exacerbation (Moderate or Severe) | up to 52 weeks
  The term from enrollment to the date of first COPD exacerbation is a duration from the start of intervention (Week0) to the date of first COPD exacerbation or death from any cause which ever comes first.
  The date of first COPD exacerbation will be assessed by the disease diary which is kept by each patient within the term of intervention.
Term from enrollment to death from any cause | up to 52 weeks
  Term from enrollment to death from any cause is a duration from the start of intervention (Week0) to death from any cause.
Frequency (the number of occurrences per year) of COPD exacerbation (All Severity and Severe only) | 52weeks
  COPD exacerbation will be assessed by the disease diary which is kept by each patient within the term of intervention.
Total St. George's respiratory questionnaire (SGRQ-C) score, and each components score (symptom score, activity score, and impact score) | at 0, 12, 24 and 52 weeks
  SGRQ-C score will be assessed by Japanese version of the SGRQ-C value sets including each components score (symptom score, activity score, and impact score).
Quality-adjusted life year (QALY) by mapping the EQ-5D-5L utility scores | at 0, 12, 24 and 52 weeks
  Quality-adjusted life year (QALY) of the subjects will be assessed by Japanese version of the EQ-5D-5L value sets including assessment of changes from baseline in the EQ-5D-5L utility index scores and visual analogue scale scores.
Total SRI (Severe Respiratory Insufficiency Questionnaire) score | at 0, 12, 24 and 52 weeks
  Total SRI score will be assessed by Japanese version of the SRI value sets.
Total PSQI-J(Japanese version of the Pittsburgh Sleep Quality Index) score | at 0, 12, 24 and 52 weeks
  Total PSQI-J score will be assessed by Japanese version of the PSQI value sets.
Dyspnea intensity: the modified medical research council (mMRC) score | 52weeks
  Dyspnea intensity will be evaluated by the modified medical research council (mMRC) score.
Arterial blood gas analysis (ABG): pH, PaO2, PaCO2, HCO3-, BE | 52weeks
  ABG will be evaluated by the blood gas analysis equipment.
Oxygen Saturation (SpO2) | 52weeks
  SpO2 will be evaluated by Pulse Oximeter.
Pulmonary functions: FVC, FEV1, FEV1% | 52weeks
  Lung function of the subjects will be assessed by the pulmonary function tests in the following indicators: vital capacity (VC, %VC), forced vital capacity (FVC, %FVC), forced expiratory volume in 1 second (FEV1, ％FEV1), FEV1/FVC.
6-minute walk test (6MWT) | at 0, 12, 24 and 52 weeks
  6MWT for the respiration rehabilitation is defined as the functional exercise capacity which is assessed by the following indicators: the distance (m), changes in pre- and post-6MWT pulse oximeter (SpO2), and post-6MWT modified borg scale.
Term from enrollment to the date of long-term (more than 1month) NPPV(Noninvasive Positive Pressure Ventilation) usage | 52weeks
  The term from the start of intervention (Week0) to the date of Long-term NPPV usage.
  Long-term NPPV usage is defined as more than 1month NPPV usage.
Flow rate(Oxygen / Total) (Arm A only) | 52weeks
  Oxygen flow rate / Total flow rate will be confirmed by the record of numerical value displayed on the device.
Total hours of myAIRVO2-use (Arm A only) | 52weeks
  Total hours of myAIRVO2-use will be confirmed by the record of numerical value displayed on the device.
Adverse events | 52weeks
  Adverse events will be determined by the latest version of MedDRA/J （Medical Dictionary for Regulatory Activities/J）at the time of Database lock.

OTHER OUTCOMES:
Correlation between frequency of COPD exacerbation (All Severity and Severe only) and amount of ABG change | 52weeks
  Amount of ABG change will be calculated by the ABG value at before and after the intervention.
Correlation between frequency of COPD exacerbation (All Severity and Severe only) and amount of SpO2 change | 52weeks
  Amount of SpO2 change will be calculated by the ABG value of before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Keisuke Tomii, MD, Ph.D., Principal Investigator — Kobe City Medical Center General Hospital
Locations (1):
- Kobe City Medical Center General Hospital, Kobe, Hyōgo, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nagata K, Horie T, Chohnabayashi N, Jinta T, Tsugitomi R, Shiraki A, Tokioka F, Kadowaki T, Watanabe A, Fukui M, Kitajima T, Sato S, Tsuda T, Kishimoto N, Kita H, Mori Y, Nakayama M, Takahashi K, Tsuboi T, Yoshida M, Hataji O, Fuke S, Kagajo M, Nishine H, Kobayashi H, Nakamura H, Okuda M, Tachibana S, Takata S, Osoreda H, Minami K, Nishimura T, Ishida T, Terada J, Takeuchi N, Kohashi Y, Inoue H, Nakagawa Y, Kikuchi T, Tomii K. Home High-Flow Nasal Cannula Oxygen Therapy for Stable Hypercapnic COPD: A Randomized Clinical Trial. Am J Respir Crit Care Med. 2022 Dec 1;206(11):1326-1335. doi: 10.1164/rccm.202201-0199OC. PMID 35771533